CLINICAL TRIAL: NCT02363842
Title: A Randomized, Controlled Trial Assessing Use of Skin IQ™ MCM Compared to Current Standard of Care for the Management of Moisture and Temperature at the Patient/Surface Interface for Prevention of Pressure Ulcer Development
Brief Title: Trial Comparing SOC +Skin IQ MCM vs SOC for Pressure Ulcer (PU)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arjohuntleigh (Industry)
Collaborators: Magellan Medical Technology Consultants, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SIQ2014-01
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer; Skin IQ MCM coverlet; Pressure redistribution surfaces
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Skin IQ™ MCM Coverlet (Experimental): Skin IQ™ MCM coverlet used over a commercially available pressure redistribution surface already in use at the participating institution to manage patients at risk for tissue breakdown
  Interventions: Device: Skin IQ™ MCM Coverlet
- Pressure redistribution surface (Active Comparator): Commercially available pressure redistribution surface already in use at participating study sites (SOC) to manage patients at risk for tissue breakdown
  Interventions: Other: Pressure redistribution surface

INTERVENTIONS:
Device: Skin IQ™ MCM Coverlet — Test article is the Skin IQ™ MCM, a Class II 510k exempt product. It is an overlay coverlet indicated to be used in conjunction with a pressure redistribution surface in order to aid in the prevention and treatment of skin breakdown and pressure ulcers for patients who require microclimate management of the skin.
  Arms: Skin IQ™ MCM Coverlet
Other: Pressure redistribution surface — Standard of Care (SOC): pressure redistribution surface already in use at the participating institution to manage patients at risk for tissue breakdown
  Arms: Pressure redistribution surface

SUMMARY:
The study is a multi-center, prospective, randomized, controlled, clinical study evaluating the effects of microclimate management using Skin IQ™ MCM coverlet placed over commercially available pressure redistribution surfaces compared to standard of care (SOC). The objective of this study is to evaluate if a commercially available pressure redistribution surface when combined with the Skin IQ™ MCM coverlet will significantly reduce pressure ulcer (PU) incidence as compared to use of a commercially available pressure redistribution surface by itself by decreasing the effects of excessive moisture and temperature at the skin and surface interface.

DETAILED DESCRIPTION:
This prospective, randomized, controlled study is designed to capture, evaluate and compare the effects of Skin IQ™ MCM coverlet placed over commercially available pressure redistribution surfaces versus commercially available pressure redistribution surface (SOC) used by itself to manage patients at risk for tissue breakdown.

Anticipation is that 160 Subjects will need to be screened and consented to achieve the desired sample size of 136 Subjects at up to 5 centers. Individual Subject, Standard Time of Observation: Up to 60 days for incidence of PU development; beyond 60 days, only hospital discharge date and disposition will be collected. The safety endpoint is the incidence of device-related serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years or older
* Deemed at risk for tissue breakdown by clinical staff via an institutional assessment protocol such as the Braden Scale, the Waterlow Scale or the Norton Scale.
* Subject, or their legal representative, is able and willing to sign an informed consent form (ICF) and willing to undergo all study related procedures.

Exclusion Criteria:

* Female Subjects who report being pregnant
* Subjects with any unstable spinal injury
* Subjects with chronic renal failure requiring dialysis at the time of enrollment
* Subjects with body mass index (BMI) > 39 as estimated at the time of enrollment
* Use of hyperbaric oxygen therapy (HBO) ≤30 days prior to screening
* Use of external warming and/or cooling devices
* Subjects who have been enrolled in this study previously
* Subjects, who in the investigator's opinion, would have any clinically significant condition that would impair the participants' ability to comply with the study procedures
* Diagnosed chronic skin disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pressure Ulcer development | Up to 60 days for incidence of Pressure Ulcer development
  Up to 60 days for incidence of Pressure Ulcer development; beyond 60 days, only hospital discharge date and disposition will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Alastair McLeod, Study Director — Arjohuntleigh, Inc.; Jean DeLeon, MD, Principal Investigator — UTSW; Susan Jones, PhD APRNCNS, Principal Investigator — Integris Baptist Hospital; Rose Ralzman, RNMScCETN(c), Principal Investigator — Rouge Valley Health System; David Mercer, Principal Investigator — UVA
Locations (4):
- United States (3):
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Texas- Southwestern, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
- Rouge Valley Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Treatment of Pressure Ulcers: Quick Reference Guide. 2009.
- [Background] Girouard K, Harrison MB, VanDenKerkof E. The symptom of pain with pressure ulcers: a review of the literature. Ostomy Wound Manage. 2008 May;54(5):30-40, 42. PMID 18493092
- [Background] Lindgren M, Unosson M, Fredrikson M, Ek AC. Immobility--a major risk factor for development of pressure ulcers among adult hospitalized patients: a prospective study. Scand J Caring Sci. 2004 Mar;18(1):57-64. doi: 10.1046/j.0283-9318.2003.00250.x. PMID 15005664
- [Background] Cullum N, McInnes E, Bell-Syer SE, Legood R. Support surfaces for pressure ulcer prevention. Cochrane Database Syst Rev. 2004;(3):CD001735. doi: 10.1002/14651858.CD001735.pub2. PMID 15266452
- [Background] Gray M, Bohacek L, Weir D, Zdanuk J. Moisture vs pressure: making sense out of perineal wounds. J Wound Ostomy Continence Nurs. 2007 Mar-Apr;34(2):134-42. doi: 10.1097/01.WON.0000264824.95860.9e. No abstract available. PMID 17413827
- [Background] Gray M. Incontinence-related skin damage: essential knowledge. Ostomy Wound Manage. 2007 Dec;53(12):28-32. PMID 18184980
- [Background] Reger SI, Ranganathan VK, Sahgal V. Support surface interface pressure, microenvironment, and the prevalence of pressure ulcers: an analysis of the literature. Ostomy Wound Manage. 2007 Oct;53(10):50-8. PMID 17978415
- [Background] Zhong W, Xing MM, Pan N, Maibach HI. Textiles and human skin, microclimate, cutaneous reactions: an overview. Cutan Ocul Toxicol. 2006;25(1):23-39. doi: 10.1080/15569520500536600. PMID 16702052
- [Background] Reger SI, Adams TC, Maklebust JA, Sahgal V. Validation test for climate control on air-loss supports. Arch Phys Med Rehabil. 2001 May;82(5):597-603. doi: 10.1053/apmr.2001.20837. PMID 11346834